CLINICAL TRIAL: NCT01593254
Title: An Open Label, Randomized (2:1) Phase IIb Study of Dasatinib Versus Imatinib in Patients With Chronic Phase Chronic Myeloid Leukemia Who Have Not Achieved an Optimal Response to 3 Months of Therapy With 400 mg Imatinib
Brief Title: Study of Dasatinib vs Imatinib in Patients With Chronic Myeloid Leukemia (CML) Who Did Not Have Favorable Response to Imatinib
Acronym: DASCERN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: ICON Clinical Research (Industry); PPD Development, LP (Industry); Molecular MD (Unknown); MultiPharma (Unknown); Q2 Solutions (Industry); Donald E. Morisky (Unknown); MD Anderson Symptom Inventory (MDASI-CML) (Unknown); OBiS, Inc (Unknown); Steering Committee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-399; 2011-006181-41 (EudraCT Number)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Imatinib (≥400 mg) (Active Comparator): Imatinib ≥400 mg tablets by mouth once daily (QD) or twice daily (BID) up to 60 months
  Interventions: Drug: Imatinib
- Arm 2: Dasatinib (100 mg) (Active Comparator): Dasatinib 100 mg tablet by mouth QD up to 60 months
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Imatinib
  Other Names: Gleevec; Glivec
  Arms: Arm 1: Imatinib (≥400 mg)
Drug: Dasatinib
  Other Names: Sprycel
  Arms: Arm 2: Dasatinib (100 mg)

SUMMARY:
The purpose of this study is to test the hypothesis that patients with CML who have not achieved optimal response after 3 months of treatment with imatinib will have a better response by switching to dasatinib compared to staying on their original imatinib regimen.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Phase (CP)-CML Ph+ patients with complete hematologic response (CHR) but without one log BCR-ABL reduction (BCR-ABL level >10% IS) 3 months of imatinib 400mg treatment. (Imatinib transient dose adjustments due to Adverse Event (AEs) are allowed with a maximum of 2 weeks interruption of treatment with imatinib (cumulative) within the 3 month period before randomization). Imatinib monotherapy must have been started within 6 months of CP-CML diagnosis (Ph + /BCR-ABL detection)
* Currently tolerating imatinib 400mg QD. Patients with prior imatinib treatment interruption or dose reductions are required to be on treatment with 400 mg imatinib for two weeks immediately prior to randomization to ensure tolerance to imatinib
* Eastern Co-Operative Group (ECOG) performance status = 0 - 2
* Adequate renal function defined as serum creatinine ≤3 times the institutional upper limit of normal (ULN)
* Adequate hepatic function defined as: total bilirubin ≤2.0 times the institutional ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the institutional ULN

Exclusion Criteria:

* Previous diagnosis of accelerated phase or blast crisis
* Subjects with clonal evolution in Ph+ cells observed in ≥2 metaphases at baseline bone marrow cytogenetic test, unless the same abnormalities were present at diagnosis. Patients with no evidence of clonal evolution, including those patients whose cytogenetic testing fails or bone marrow aspiration is a dry tap at 3 months, are eligible for the study
* Subjects with less than CHR after 3 months of imatinib treatment or lost CHR after initial achievement
* Documented T315I/A, F317L, or V299L mutations (if already available - not required for screening)
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (101):
- United States (21):
  - Local Institution - 0004, Anaheim, California
  - Local Institution - 0006, Fontana, California
  - University Of Southern California University Hospital, Los Angeles, California
  - Local Institution - 0110, Roseville, California
  - Local Institution - 0112, San Jose, California
  - Local Institution - 0009, Vallejo, California
  - Local Institution - 0078, Whittier, California
  - Local Institution - 0089, Southington, Connecticut
  - Northwestern University, Evanston, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northern Indiana Cancer Research Consortium, Crown Point, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - University Of Iowa, Iowa City, Iowa
  - Local Institution - 0010, Rochester, Minnesota
  - Local Institution - 0002, Cincinnati, Ohio
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Local Institution - 0001, Nashville, Tennessee
  - Michael E Debakey VAMC, Houston, Texas
  - Institute of Oncology Hematology Biomedical Research, Laredo, Texas
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Local Institution - 0005, Milwaukee, Wisconsin
- Argentina (6):
  - Local Institution - 0093, La Plata, Buenos Aires
  - Local Institution - 0080, Ramos Mejía, Buenos Aires
  - Local Institution - 0049, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0051, Buenos Aires
  - Local Institution - 0057, Buenos Aires
  - Local Institution - 0100, Corrientes
- Austria (6):
  - Local Institution - 0026, Innsbruck, Tyrol
  - Local Institution - 0022, Wels, Upper Austria
  - Local Institution, Fürstenfeld
  - Local Institution - 0043, Graz
  - Local Institution - 0024, Linz
  - Local Institution - 0023, Vienna
- Belgium (3):
  - Local Institution - 0065, Bruges
  - Local Institution - 0099, Merksem
  - Local Institution, Yvoir
- Brazil (8):
  - Local Institution - 0083, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution - 0063, Campinas, São Paulo
  - Local Institution, Ribeirão Preto, São Paulo
  - Local Institution - 0059, São Paulo, São Paulo
  - Local Institution - 0062, Rio de Janeiro
  - Local Institution - 0058, Rio de Janeiro
  - Local Institution - 0111, Rio de Janeiro
- Local Institution - 0020, Saint John, New Brunswick, Canada
- China (18):
  - Local Institution - 0071, Beijing, Beijing Municipality
  - Local Institution - 0086, Beijing, Beijing Municipality
  - Local Institution - 0070, Fuzhou, Fujian
  - Local Institution - 0103, Shenzhen, Guandong
  - Local Institution - 0082, Guangzhou, Guangdong
  - Local Institution - 0074, Guangzhou, Guangdong
  - Local Institution - 0084, Haerbin, Heilongjiang
  - Local Institution - 0102, Wuhan, Hubei
  - Local Institution - 0073, Nanjing, Jiangsu
  - Local Institution - 0077, Suzhou, Jiangsu
  - Local Institution - 0094, Shenyang, Liaoning
  - Local Institution - 0088, Xi'an, Shan3xi
  - Local Institution - 0101, Jinan, Shandong
  - Local Institution - 0075, Chengdu, Sichuan
  - Local Institution - 0069, Tianjin, Tianjin Municipality
  - Local Institution - 0072, Hangzhou
  - Local Institution - 0076, Shanghai
  - Local Institution - 0096, Wuhan
- Czechia (5):
  - Local Institution - 0032, Brno, Czech Republic
  - Local Institution, Hradec Králové
  - Local Institution, Olomouc
  - Local Institution, Prague
  - Local Institution - 0067, Prague
- France (5):
  - Local Institution - 0045, Le Chesnay
  - Local Institution - 0041, Lille
  - Local Institution, Nantes
  - Local Institution, Pierre-Bénite
  - Local Institution - 0038, Vandœuvre-lès-Nancy
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution - 0104, Szeged
- Italy (10):
  - Local Institution - 0106, Brescia, Province Of Brescia
  - Local Institution, Bari
  - Local Institution, Bologna
  - Local Institution, Catania
  - Local Institution - 0027, Florence
  - Local Institution - 0046, Monza
  - Local Institution, Napoli
  - Local Institution - 0025, Orbassano
  - Local Institution - 0021, Roma
  - Local Institution - 0033, Rome
- Poland (4):
  - Local Institution - 0048, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0047, Gdansk
  - Local Institution - 0098, Katowice
  - Local Institution - 0064, Warsaw
- South Korea (3):
  - Local Institution - 0039, Seoul
  - Local Institution - 0050, Seoul
  - Local Institution - 0040, Seoul
- Spain (6):
  - Local Institution - 0017, A Couruna
  - Local Institution - 0018, L'Hospitalet Del Llobregat
  - Local Institution - 0015, Las Palmas de Gran Canaria
  - Local Institution - 0012, Madrid
  - Local Institution - 0013, Salamanca
  - Local Institution - 0011, Toledo
- Thailand (3):
  - Local Institution - 0055, Muang, Chiang Mai
  - Local Institution, Bangkok
  - Local Institution - 0052, Khon Kaen

REFERENCES:
- [Derived] Cortes JE, Jiang Q, Wang J, Weng J, Zhu H, Liu X, Hochhaus A, Kim DW, Radich J, Savona M, Martin-Regueira P, Sy O, Gurnani R, Saglio G. Dasatinib vs. imatinib in patients with chronic myeloid leukemia in chronic phase (CML-CP) who have not achieved an optimal response to 3 months of imatinib therapy: the DASCERN randomized study. Leukemia. 2020 Aug;34(8):2064-2073. doi: 10.1038/s41375-020-0805-1. Epub 2020 Apr 7. PMID 32265500
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 260 participants treated
Period: Overall Study
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Started (Started = Started Treatment Period) | 86 | 174
Crossed Over to Dasatinib | 46 | 0
Completed (Completed = Continuing in Treatment Period) | 0 | 0
Not Completed | 86 | 174
Not completed — Disease progression | 2 | 7
Not completed — Study drug toxicity | 6 | 20
Not completed — Death | 3 | 3
Not completed — AE unrelated to study drug | 0 | 1
Not completed — participant request to discontinue study treatment | 1 | 3
Not completed — participant withdrew consent | 0 | 9
Not completed — lost to follow up | 1 | 6
Not completed — maximum clinical benefit | 1 | 2
Not completed — Poor/non compliance | 1 | 1
Not completed — Pregnancy | 0 | 3
Not completed — participant no longer meets study criteria | 1 | 1
Not completed — Admin reason by sponsor | 7 | 3
Not completed — Imatinib treatment failure | 2 | 0
Not completed — Other Reasons | 61 | 115

BASELINE CHARACTERISTICS:
Population: All Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 2: Dasatinib (100 mg) | Arm 1: Imatinib (≥400 mg) | Total
Number analyzed (Participants) | 174 | 86 | 260
Age, Continuous [Median (Full Range); unit: years] — Population: All Randomized Participants
  years | 35.0 [18 to 82] | 39.5 [18 to 73] | 37.0 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Randomized Participants
  Participants
    Female | 41 | 16 | 57
    Male | 133 | 70 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Randomized Participants
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 174 | 86 | 260
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Randomized Participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 127 | 63 | 190
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 3 | 7
    White | 36 | 15 | 51
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Major Molecular Response (MMR) After 12 Months of CML Treatment
Description: Major Molecular Response, is defined as a 3-log reduction in BCR-ABL transcripts from the standardized baseline, which represents 100% on the international scale, so a 3-log reduction is fixed at 0.1% for MMR; N/A = not applicable. 95% CI is Clopper-Pearson(Exact) two-sided 95% confidence intervals.
  P-value is based on Cochran-Mantel-Haenszel (CMH) test stratified by Sokal score(high, intermediate, low, and unknown) and time between 3 month molecular analysis and randomization (<=4 weeks vs >4 weeks).
Time Frame: At 12 months after Day 1 initiation of 1st line treatment with imatinib or imatinib at any dose, after less than optimal response to first-line imatinib.
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Number analyzed (Participants) | 86 | 174
Percentage of Patients | 12.8 [6.6 to 21.7] | 28.7 [22.1 to 36.1]
Statistical Analysis 1: Comparison: Arm 1: Imatinib (≥400 mg) vs Arm 2: Dasatinib (100 mg); Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel

2. Secondary Outcome: Median Time to Major Molecular Response (MMR)
Description: Median Time to Major Molecular Response (MMR) is the time between randomization date and first date that MMR (or MR4.5) criteria are satisfied. Participants who do not achieve MMR (or MR4.5) will be censored.
  Major Molecular Response, is defined as a 3-log reduction in BCR-ABL transcripts from the standardized baseline, which represents 100% on the international scale, so a 3-log reduction is fixed at 0.1% for MMR.
Time Frame: From randomization to study completion. Approximately 115 months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Number analyzed (Participants) | 86 | 174
Months | 19.7 [14.2 to 26.4] | 13.9 [11.6 to 17.6]

3. Secondary Outcome: Time to Molecular Response (MR)^4.5
Description: Time to Molecular Response (MR)^4.5 is the time between randomization date and first date that MMR (or MR4.5) criteria are satisfied. Participants who do not achieve MMR (or MR4.5) will be censored.
  MR4.5 is defined as a 4.5-log reduction in BCR-ABL transcript from the standardized baseline (0.0032% IS, either detectable disease <= 0.0032% BCR-ABL (IS) or undetectable disease in cDNA (in same volume used for BCR-ABL) with >= 32,000 ABL transcripts.
Time Frame: From randomization to study completion. Approximately 115 months
Population: All Randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Number analyzed (Participants) | 86 | 174
Months | 67.7 [55.9 to NA] — insufficient number of participants with events to calculate via KM methodology | 74.5 [67.1 to 91.8]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the time from randomization date to progression date or death date, whichever occurs first. Participants who neither progress nor die will be censored.
  Progression is defined as the following, meeting the criteria for accelerated or blast crisis CML are met at any time or death from any cause during treatment.
  Accelerated phase of CML:
  * The presence of ≥15%, but < 30% blasts in the blood or bone marrow
  * At least 30% blasts plus promyelocytes in the blood or bone marrow
  * At least 20% peripheral basophils
  * Thrombocytopenia (fewer than 100,000 platelets/mm3) unrelated to treatment.
  Blast phase of CML
  * At least 30% blasts in the blood or bone marrow
  * Extramedullary involvement (e.g., chloromas), but not hepatosplenomegaly
Time Frame: From randomization to study completion. Approximately 115 months
Population: All randomized participants with a progression event
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Number analyzed (Participants) | 7 | 15
Months | NA [89.3 to NA] — insufficient number of participants with events to calculate via KM methodology | NA [NA to NA] — insufficient number of participants with events to calculate via KM methodology

5. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from randomization date to death date. Participants who have not died will be censored on the last date they are known to be alive.
Time Frame: From randomization to study completion. Approximately 115 months
Population: All randomized participants who died
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Imatinib (≥400 mg) | Arm 2: Dasatinib (100 mg)
Number analyzed (Participants) | 5 | 11
Months | NA [89.3 to NA] — insufficient number of participants with events to calculate via KM methodology | NA [NA to NA] — insufficient number of participants with events to calculate via KM methodology

ADVERSE EVENTS:
Time Frame: From first dose date up to 30 days after last dose of study therapy. Assessed from Sept. 2012 to Nov. 2017 (approximately 62 months) All cause mortality is from the time of randomization to the end of study. Approximately 115 months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Arm 1: Imatinib: Imatinib ≥400 mg tablets by mouth once daily (QD) or twice daily (BID) up to 60 months.
- Arm 2: Dasatinib: Dasatinib 100 mg tablet by mouth QD up to 60 months
- Dasatinib After Crossover From Imatinib: Dasatinib 100 mg tablet by mouth QD
Arm/Group | Arm 1: Imatinib | Arm 2: Dasatinib | Dasatinib After Crossover From Imatinib
All-Cause Mortality (participants affected / at risk) | 1/86 | 11/174 | 4/46
Serious Adverse Events (participants affected / at risk) | 11/86 | 48/171 | 8/46
Other Adverse Events (participants affected / at risk) | 68/86 | 159/171 | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Imatinib (N=86) | Arm 2: Dasatinib (N=171) | Dasatinib After Crossover From Imatinib (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Anal abscess (Infections and infestations) | 0 | 2 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Complicated appendicitis (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 6
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Tuberculosis of central nervous system (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Paternal exposure timing unspecified (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Imatinib (N=86) | Arm 2: Dasatinib (N=171) | Dasatinib After Crossover From Imatinib (N=46)
Anaemia (Blood and lymphatic system disorders) | 20 | 53 | 15
Leukopenia (Blood and lymphatic system disorders) | 8 | 17 | 8
Neutropenia (Blood and lymphatic system disorders) | 20 | 42 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 40 | 10
Pericardial effusion (Cardiac disorders) | 0 | 9 | 4
Eyelid oedema (Eye disorders) | 8 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 14 | 4
Diarrhoea (Gastrointestinal disorders) | 11 | 33 | 8
Nausea (Gastrointestinal disorders) | 9 | 17 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9 | 0
Asthenia (General disorders) | 2 | 11 | 2
Fatigue (General disorders) | 7 | 9 | 0
Pyrexia (General disorders) | 3 | 21 | 10
Bronchitis (Infections and infestations) | 5 | 7 | 1
Influenza (Infections and infestations) | 1 | 10 | 0
Nasopharyngitis (Infections and infestations) | 6 | 16 | 4
Upper respiratory tract infection (Infections and infestations) | 13 | 29 | 12
Alanine aminotransferase increased (Investigations) | 8 | 14 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 15 | 4
Blood bilirubin increased (Investigations) | 4 | 14 | 2
Blood cholesterol increased (Investigations) | 1 | 12 | 1
Blood creatine phosphokinase increased (Investigations) | 11 | 19 | 4
Blood lactate dehydrogenase increased (Investigations) | 2 | 14 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 11 | 1
Haemoglobin decreased (Investigations) | 3 | 11 | 5
High density lipoprotein decreased (Investigations) | 2 | 10 | 1
Low density lipoprotein increased (Investigations) | 0 | 9 | 0
Neutrophil count decreased (Investigations) | 13 | 26 | 13
Platelet count decreased (Investigations) | 19 | 36 | 12
Weight increased (Investigations) | 2 | 5 | 3
White blood cell count decreased (Investigations) | 15 | 26 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 12 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 14 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 9 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 18 | 27 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 11 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 10 | 1
Dizziness (Nervous system disorders) | 6 | 11 | 1
Headache (Nervous system disorders) | 3 | 40 | 6
Insomnia (Psychiatric disorders) | 7 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 24 | 9
Rash (Skin and subcutaneous tissue disorders) | 8 | 21 | 3
Hypertension (Vascular disorders) | 5 | 11 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT01593254/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT01593254/SAP_001.pdf